CLINICAL TRIAL: NCT05408169
Title: Increasing Uptake of Faecal Immunochemical Test (FIT) Bowel Screening: Trial of Providing a Suggested Deadline for FIT Kit Return and a Planning Sheet
Brief Title: Increasing Uptake of Bowel Screening
Acronym: TEMPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); NHS Tayside (Other Government); University of Cambridge (Other); University of St Andrews (Other); University of Stirling (Other); University of Dundee (Other); Chief Scientist Office of the Scottish Government (Other Government); Cancer Research UK (Other)
Responsible Party: Principal Investigator, Katie Robb, Professor of Behavioural Science and Health, University of Glasgow
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Health Services Research
Other Study IDs: GN19GA165
Record Dates: First submitted 2022-04-29; First posted 2022-06-07 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Cancer
Keywords: Early Detection of Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Control (No Intervention)
- 1-week deadline, no planning sheet (Experimental)
  Interventions: Behavioral: Suggested deadline for return of screening test
- 2-week deadline, no planning sheet (Experimental)
  Interventions: Behavioral: Suggested deadline for return of screening test
- 4-week deadline, no planning sheet (Experimental)
  Interventions: Behavioral: Suggested deadline for return of screening test
- No deadline, with planning sheet (Experimental)
  Interventions: Behavioral: Planning sheet
- 1-week deadline, with planning sheet (Experimental)
  Interventions: Behavioral: Suggested deadline for return of screening test; Behavioral: Planning sheet
- 2-week deadline, with planning sheet (Experimental)
  Interventions: Behavioral: Suggested deadline for return of screening test; Behavioral: Planning sheet
- 4-week deadline, with planning sheet (Experimental)
  Interventions: Behavioral: Suggested deadline for return of screening test; Behavioral: Planning sheet

INTERVENTIONS:
Behavioral: Suggested deadline for return of screening test — A screening invitation letter modified to state, highlighted in yellow: "Please return your kit within [X] weeks (by [DD.MM.YYYY]) or as soon as possible."
  Arms: 1-week deadline, no planning sheet; 1-week deadline, with planning sheet; 2-week deadline, no planning sheet; 2-week deadline, with planning sheet; 4-week deadline, no planning sheet; 4-week deadline, with planning sheet
Behavioral: Planning sheet — A planning tool presented on a separate single sheet of paper inserted into the screening invitation envelope. The colour illustrated tool prompts participants to identify concerns they have with using the bowel screening kit and to link them to a tip to help them overcome this concern.
  Other Names: Volitional help sheet
  Arms: 1-week deadline, with planning sheet; 2-week deadline, with planning sheet; 4-week deadline, with planning sheet; No deadline, with planning sheet

SUMMARY:
Bowel cancer is the second biggest cancer killer in the UK, accounting for over 16,000 deaths per year. Screening can reduce deaths from bowel cancer if the people invited participate. The challenge is that high uptake of bowel screening is hard to achieve, and remains persistently below 65%.

The faecal immunochemical test (FIT) is the most widely used bowel screening test worldwide.

In the UK, FIT kits are mailed to people's homes without guidance on when the kit should be returned and only brief instruction on how to use it. Some people have said that even though they intend to complete and return the kit, they often forget or put off doing it.

Two approaches are proposed to addressing this issue: i) providing a suggested deadline for FIT return, because it is known from breast and cervical cancer screening that giving people an appointment time increases uptake compared to an open invitation, and ii) planning sheets, that have been found to help people act on their intentions in other health contexts.

This trial aims to evaluate the impact of providing a suggested deadline and a planning sheet on the return of FIT bowel screening kits.

The trial is integrated within the Scottish Bowel Screening Programme. The investigators will randomly allocate 40,000 consecutive people that are due to be sent a FIT kit to one of eight groups:

(i) control group (no deadline, no planning sheet), (ii) intervention group (1-week deadline, no planning sheet), (iii) intervention group (2-week deadline, no planning sheet), (iv) intervention group (4-week deadline, no planning sheet), (v) intervention group (no deadline, with planning sheet), (vi) intervention group (1-week deadline, with planning sheet), (vii) intervention group (2-week deadline, with planning sheet), (viii) intervention group (4-week deadline, with planning sheet).

It will then be examined if having a suggested deadline and a planning sheet affects how many people send back their completed FIT kit. It will also be examined if the deadline length makes a difference and whether having both a deadline and a planning sheet affects the number of people returning their kit.

Finally, the cognitive and behavioural mechanisms underlying any intervention effects will be assessed and the acceptability of the interventions explored, using questionnaires and in-depth interviews.

ELIGIBILITY:
Inclusion Criteria:

* 50-74 years
* Registered with a Community Health Index number in Scotland
* More than 2 years since last bowel screening invitation

Exclusion Criteria:

* Has self-excluded from Scottish Bowel Screening Programme
* Not sent a screening kit by the Scottish Bowel Screening Programme

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40000 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of screening tests returned to the central laboratory and successfully processed providing an adequate result. | 3 months

SECONDARY OUTCOMES:
Number of screening tests returned to the central laboratory | 3 months
Number of screening tests returned to the central laboratory within suggested deadline | 1/2/4 weeks
Number of screening tests returned to the central laboratory by area-level deprivation | 3 months
Cognitive and behavioural mechanisms | 3 months
  A questionnaire designed to assess mechanisms, e.g. action and coping planning, using items adapted for the bowel screening context.
Acceptability of interventions (quantitative) | 3 months
  The Acceptability Questionnaire
Acceptability of interventions (qualitative) | 3-8 months
  Analysis of in-depth semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Robb, Principal Investigator — University of Glasgow
Locations (1):
- Scottish Bowel Screening Centre, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Outcomes 1-4: Details of the dataset and work arising from it will be available from the Robertson Centre for Biostatistics Analytical Platform at the University of Glasgow. The dataset will be archived on live servers within the facility. Use of anonymised data within research is given for the specified project purpose, future use is permitted but would require permission from LPAC and the Caldicott Guardian.
  Outcomes 5-6: Quantitative data (SPSS files with metadata) and qualitative data (stored as MSword transcripts with metadata) will be deposited in Enlighten: Research Data, the University of Glasgow's institutional data repository. Data in the repository will be stored in accordance with funder and University data policies. Files will be given a Digital Object Identifier (DOI) and the associated metadata will be listed in the University of Glasgow Research Data Registry and the DataCite metadata store.
Time Frame: Outcomes 1-4: 5 years post completion and data then moved to off-line storage.
  Outcomes 5-6: 10 years from date of deposition in the first instance, with extensions applied to datasets which are subsequently accessed.
Access Criteria: Outcomes 1-4: There is no requirement for a data sharing agreement with the research team and no restrictions on data sharing. Any research group can approach and request permission to use datasets.
  Outcomes 5-6: Data made public at the time of publication.

REFERENCES:
- [Derived] Robb KA, Young B, Murphy MK, Duklas P, McConnachie A, Hollands GJ, McCowan C, Macdonald S, O'Carroll RE, O'Connor RC, Steele RJC. Behavioural interventions to increase uptake of FIT colorectal screening in Scotland (TEMPO): a nationwide, eight-arm, factorial, randomised controlled trial. Lancet. 2025 Mar 29;405(10484):1081-1092. doi: 10.1016/S0140-6736(24)02813-7. Epub 2025 Mar 12. PMID 40088914
- [Derived] Robb KA, Kotzur M, Young B, McCowan C, Hollands GJ, Irvine A, Macdonald S, McConnachie A, O'Carroll RE, O'Connor RC, Steele RJC. Increasing uptake of FIT colorectal screening: protocol for the TEMPO randomised controlled trial testing a suggested deadline and a planning tool. BMJ Open. 2023 May 18;13(5):e066136. doi: 10.1136/bmjopen-2022-066136. PMID 37202130